CLINICAL TRIAL: NCT06528314
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Efruxifermin in Subjects With Compensated Cirrohosis Due to NASH/MASH
Brief Title: A Study Evaluating Efruxifermin in Subjects With Compensated Cirrhosis Due to NASH/MASH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akero Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK-US-001-0106
Record Dates: First submitted 2024-06-28; First posted 2024-07-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; MASH - Metabolic Dysfunction-Associated Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EFX 50 mg (Experimental)
  Interventions: Drug: Efruxifermin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efruxifermin — Administered by subcutaneous injection
  Arms: EFX 50 mg
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a multi-center evaluation of efruxifermin (EFX) in a randomized, double-blind, placebo-controlled study in subjects with compensated cirrhosis due to NASH/MASH.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Biopsy proven compensated cirrhosis (fibrosis stage 4) due to NASH/MASH
* Cohort 2: Biopsy proven or non-invasively diagnosed compensated cirrhosis (fibrosis stage 4) due to NASH/MASH

Exclusion Criteria:

* Other causes of liver disease based on medical history and/or liver histology and/or central laboratory results
* Type 1 diabetes or unstable Type 2 diabetes
* Any current or prior history of decompensated liver disease

Other inclusion and exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to first occurrence of disease progression as measured by composite of protocol-specified clinical events | 5 years
Cohort 1 only: ≥ 1 stage improvement in fibrosis and no worsening of steatohepatitis | 96 Weeks
  Based on NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)

SECONDARY OUTCOMES:
Change from baseline of non-invasive markers of liver fibrosis | 96 Weeks
  ELF (scale of 6.7 to 11.3 with higher scores indicative of increased fibrosis)
Change from baseline of non-invasive markers of liver fibrosis | 96 Weeks
  Pro-C3 (ug/L)
Change from baseline of non-invasive markers of liver fibrosis | 96 Weeks
  Liver stiffness assessed by transient elastography (FibroScan®) (kPa)
Change from baseline of non-invasive markers of liver fibrosis | 96 Weeks
  FAST score (varied on a scale from 0 to 1, with the patients being classified as having low [<0.35], intermediate [0.35-0.67], or higher [>0.67] probability of having significant inflammatory activity and fibrosis)
Change from baseline of markers of liver injury | 96 Weeks
  ALT (U/L) and AST (U/L)
Change from baseline of lipoproteins | 96 Weeks
  Total cholesterol (mg/dL), Triglycerides (mg/dL), HDL-C (mg/dL), Non-HDL-C (mg/dL), and LDL-C (mg/dL)
Change from baseline of markers of insulin sensitivity and glycemic control | 96 Weeks
  HbA1c (%)
Change from baseline of markers of insulin sensitivity and glycemic control | 96 Weeks
  C-Peptide (ng/mL)
Change from baseline of markers of insulin sensitivity and glycemic control | 96 Weeks
  Adiponectin (mg/L)
Change from baseline of markers of insulin sensitivity and glycemic control | 96 Weeks
  Insulin (mIU/L)
Change from baseline of markers of insulin sensitivity and glycemic control | 96 Weeks
  HOMA-IR (≥ 2.5 indicates insulin resistance)
Change from baseline of body weight (kg) | 96 Weeks
To assess the safety and tolerability of EFX through the reporting of extent of exposure (weeks) | 96 Weeks
To assess the safety and tolerability of EFX through the reporting of adverse events (frequency of events) | 96 Weeks
To assess the safety and tolerability of EFX through the reporting of adverse events (severity of events) | 96 Weeks
Number of participants with abnormal laboratory tests results, abnormal ECGs, abnormal ultrasounds, abnormal vital sign assessments | 96 Weeks
Cohort 1 only: ≥ 1 stage improvement in fibrosis and no worsening of steatohepatitis | 5 Years
  Based on NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)
Cohort 1 only: ≥ 1 stage improvement in fibrosis | 96 Weeks, 5 Years
  Based on NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)
Cohort 1 only: Resolution of NASH/MASH | 96 Weeks, 5 Years
  Based on NAS (scored by 0-1 for steatosis, 0-3 for inflammation, and 0-2 for ballooning)
Cohort 1 only: Resolution of NASH/MASH and a ≥ 1 stage improvement in fibrosis | 96 Weeks, 5 Years
  Based on NAS (scored by 0-1 for steatosis, 0-3 for inflammation, and 0-2 for ballooning) and NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)

CONTACTS AND LOCATIONS:
Locations (258):
- United States (133):
  - Akero Clinical Study Site, Birmingham, Alabama
  - Akero Clinical Study Site, Dothan, Alabama
  - Akero Clinical Study Site, Chandler, Arizona
  - Akero Clinical Study Site, Flagstaff, Arizona
  - Akero Clinical Study Site, Peoria, Arizona
  - Akero Clinical Study Site, Scottsdale, Arizona
  - Akero Clinical Study Site, Tucson, Arizona
  - Akero Clinical Study Site, Conway, Arkansas
  - Akero Clinical Study Site, Jonesboro, Arkansas
  - Akero Clinical Study Site, Little Rock, Arkansas
  - Akero Clinical Study Site, North Little Rock, Arkansas
  - Akero Clinical Study Site, Coronado, California
  - Akero Clinical Study Site, Escondido, California
  - Akero Clinical Study Site, Folsom, California
  - Akero Clinical Study Site, Lancaster, California
  - Akero Clinical Study Site, Long Beach, California
  - Akero Clinical Study Site, Los Angeles, California
  - Akero Clinical Study Site, Newport Beach, California
  - Akero Clinical Study Site, Orange, California
  - Akero Clinical Study Site, Pasadena, California
  - Akero Clinical Study Site, Redwood City, California
  - Akero Clinical Study Site, San Francisco, California
  - Akero Clinical Study Site, San Jose, California
  - Akero Clinical Study Site, Aurora, Colorado
  - Akero Clinical Study Site, Colorado Springs, Colorado
  - Akero Clinical Study Site, Englewood, Colorado
  - Akero Clinical Study Site, New Haven, Connecticut
  - Akero Clinical Study Site, Washington D.C., District of Columbia
  - Akero Clinical Study Site, Bradenton, Florida
  - Akero Clinical Study Site, Brandon, Florida
  - Akero Clinical Study Site, Cutler Bay, Florida
  - Akero Clinical Study Site, Doral, Florida
  - Akero Clinical Study Site, Fort Myers, Florida
  - Akero Clinical Study Site, Hialeah Gardens, Florida
  - Akero Clinical Study Site, Inverness, Florida
  - Akero Clinical Study Site, Lakewood Rch, Florida
  - Akero Clinical Study Site, Largo, Florida
  - Akero Clinical Study Site, Lehigh Acres, Florida
  - Akero Clinical Study Site, Margate, Florida
  - Akero Clinical Study Site, Miami, Florida
  - Akero Clinical Study Site, Miami Gardens, Florida
  - Akero Clinical Study Site, Naples, Florida
  - Akero Clinical Study Site, New Port Richey, Florida
  - Akero Clinical Study Site, Ocala, Florida
  - Akero Clinical Study Site, Orlando, Florida
  - Akero Clinical Study Site, Pembroke Pines, Florida
  - Akero Clinical Study Site, Riverview, Florida
  - Akero Clinical Study Site, Sarasota, Florida
  - Akero Clinical Study Site, Temple Terrace, Florida
  - Akero Clinical Study Site, Venice, Florida
  - Akero Clinical Study Site, Weston, Florida
  - Akero Clinical Study Site, Zephyrhills, Florida
  - Akero Clinical Study Site, Atlanta, Georgia
  - Akero Clinical Study Site, Gainesville, Georgia
  - Akero Clinical Study Site, Marietta, Georgia
  - Akero Clinical Study Site, Snellville, Georgia
  - Akero Clinical Study Site, Chicago, Illinois
  - Akero Clinical Study Site, Hammond, Indiana
  - Akero Clinical Study Site, Indianapolis, Indiana
  - Akero Clinical Study Site, South Bend, Indiana
  - Akero Clinical Study Site, West Des Moines, Iowa
  - Akero Clinical Study Site, Topeka, Kansas
  - Akero Clinical Study Site, Louisville, Kentucky
  - Akero Clinical Study Site, Bastrop, Louisiana
  - Akero Clinical Study Site, Covington, Louisiana
  - Akero Clinical Study Site, Houma, Louisiana
  - Akero Clinical Study Site, Lafayette, Louisiana
  - Akero Clinical Study Site, Marrero, Louisiana
  - Akero Clinical Study Site, Metairie, Louisiana
  - Akero Clinical Study Site, Shreveport, Louisiana
  - Akero Clinical Study Site, West Monroe, Louisiana
  - Akero Clinical Study Site, Baltimore, Maryland
  - Akero Clinical Study Site, Bethesda, Maryland
  - Akero Clinical Study Site, South Dartmouth, Massachusetts
  - Akero Clinical Study Site, Clinton Township, Michigan
  - Akero Clinical Study Site, Novi, Michigan
  - Akero Clinical Study Site, Southfield, Michigan
  - Akero Clinical Study Site, Rochester, Minnesota
  - Akero Clinical Study Site, Flowood, Mississippi
  - Akero Clinical Study Site, Columbia, Missouri
  - Akero Clinical Study Site, Kansas City, Missouri
  - Akero Clinical Study Site, St Louis, Missouri
  - Akero Clinical Study Site, Las Vegas, Nevada
  - Akero Clinical Study Site, Jackson, New Jersey
  - Akero Clinical Study Site, Somers Point, New Jersey
  - Akero Clinical Study Site, Sparta, New Jersey
  - Akero Clinical Study Site, Buffalo, New York
  - Akero Clinical Study Site, Manhasset, New York
  - Akero Clinical Study Site, New York, New York
  - Akero Clinical Study Site, Rochester, New York
  - Akero Clinical Study Site, Chapel Hill, North Carolina
  - Akero Clinical Study Site, Charlotte, North Carolina
  - Akero Clinical Study Site, Durham, North Carolina
  - Akero Clinical Study Site, Fayetteville, North Carolina
  - Akero Clinical Study Site, Morehead City, North Carolina
  - Akero Clinical Study Site, Raleigh, North Carolina
  - Akero Clinical Study Site, Statesville, North Carolina
  - Akero Clinical Study Site, Akron, Ohio
  - Akero Clinical Study Site, Springboro, Ohio
  - Akero Clinical Study Site, Westlake, Ohio
  - Akero Clinical Study Site, Hershey, Pennsylvania
  - Akero Clinical Study Site, Philadelphia, Pennsylvania
  - Akero Clinical Study Site, Pittsburgh, Pennsylvania
  - Akero Clinical Study Site, Charleston, South Carolina
  - Akero Clinical Study Site, Columbia, South Carolina
  - Akero Clinical Study Site, Summerville, South Carolina
  - Akero Clinical Study Site, Clarksville, Tennessee
  - Akero Clinical Study Site, Hermitage, Tennessee
  - Akero Clinical Study Site, Nashville, Tennessee
  - Akero Clinical Study Site, Amarillo, Texas
  - Akero Clinical Study Site, Austin, Texas
  - Akero Clinical Study Site, Bellaire, Texas
  - Akero Clinical Study Site, Brownsville, Texas
  - Akero Clinical Study Site, Corpus Christi, Texas
  - Akero Clinical Study Site, Dallas, Texas
  - Akero Clinical Study Site, Denison, Texas
  - Akero Clinical Study Site, Edinburg, Texas
  - Akero Clinical Study Site, Fort Sam Houston, Texas
  - Akero Clinical Study Site, Fort Worth, Texas
  - Akero Clinical Study Site, Garland, Texas
  - Akero Clinical Study Site, Houston, Texas
  - Akero Clinical Study Site, Pasadena, Texas
  - Akero Clinical Study Site, Pharr, Texas
  - Akero Clinical Study Site, San Antonio, Texas
  - Akero Clinical Study Site, Sugar Land, Texas
  - Akero Clinical Study Site, Waco, Texas
  - Akero Clinical Study Site, Webster, Texas
  - Akero Clinical Study Site, Wichita Falls, Texas
  - Akero Clinical Study Site, Norfolk, Virginia
  - Akero Clinical Study Site, Richmond, Virginia
  - Akero Clinical Study Site, Roanoke, Virginia
  - Akero Clinical Study Site, Seattle, Washington
  - Akero Clinical Study Site, Madison, Wisconsin
- Argentina (6):
  - Akero Clinical Study Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Akero Clinical Study Site, La Plata, Buenos Aires
  - Akero Clinical Study Site, Ramos Mejía, Buenos Aires
  - Akero Clinical Study Site, Buenos Aires, Distrito Federal
  - Akero Clinical Study Site, Rosario, Sante Fe
  - Akero Clinical Study Site, Buenos Aires
- Australia (13):
  - Akero Clinical Study Site, Broadmeadow, New South Wales
  - Akero Clinical Study Site, Liverpool, New South Wales
  - Akero Clinical Study Site, Westmead, New South Wales
  - Akero Clinical Study Site, Herston, Queensland
  - Akero Clinical Study Site, Adelaide, South Australia
  - Akero Clinical Study Site, Box Hill, Victoria
  - Akero Clinical Study Site, Clayton, Victoria
  - Akero Clinical Study Site, Epping, Victoria
  - Akero Clinical Study Site, Heidelberg, Victoria
  - Akero Clinical Study Site, Melbourne, Victoria
  - Akero Clinical Study Site, Murdoch, Western Australia
  - Akero Clinical Study Site, Nedlands, Western Australia
  - Akero Clinical Study Site, Perth, Western Australia
- Brazil (4):
  - Akero Clinical Study Site, Brasília, Federal District
  - Akero Clinical Study Site, Goiânia, Goiás
  - Akero Clinical Study Site, Belo Horizonte, Minas Gerais
  - Akero Clinical Study Site, Porto Alegre, Rio Grande do Sul
- Canada (5):
  - Akero Clinical Study Site, Edmonton, Alberta
  - Akero Clinical Study Site, Toronto, Ontario
  - Akero Clinical Study Site, Vaughan, Ontario
  - Akero Clinical Study Site, Montreal, Quebec
  - Akero Clinical Study Site, Terrebonne, Quebec
- Chile (3):
  - Akero Clinical Study Site, La Serena, Coquimbo Region
  - Akero Clinical Study Site, Las Condes, Santiago Metropolitan
  - Akero Clinical Study Site, Santiago, Santiago Metropolitan
- France (14):
  - Akero Clinical Study Site, Strasbourg, Bas-Rhin
  - Akero Clinical Study Site, Limoges, Haute-Vienne
  - Akero Clinical Study Site, Lille, Hauts-de-France
  - Akero Clinical Study Site, Clichy, Hauts-de-Seine
  - Akero Clinical Study Site, Vandœuvre-lès-Nancy, Lorraine
  - Akero Clinical Study Site, Angers, Maine-et-Loire
  - Akero Clinical Study Site, Toulouse, Occitanie
  - Akero Clinical Study Site, Marseille, Provence-Alpes-Côte d'Azur Region
  - Akero Clinical Study Site, Montpellier Cedex 5, Provence-Alpes-Côte d'Azur Region
  - Akero Clinical Study Site, Nice, Provence-Alpes-Côte d'Azur Region
  - Akero Clinical Study Site, Lyon, Rhône
  - Akero Clinical Study Site, Créteil, Val-de-Marne
  - Akero Clinical Study Site, Le Chesnay, Île-de-France Region
  - Akero Clinical Study Site, Paris, Île-de-France Region
- Germany (5):
  - Akero Clinical Study Site, Frankfurt am Main, Hesse
  - Akero Clinical Study Site, Homburg, Saarland
  - Akero Clinical Study Site, Leipzig, Saxony
  - Akero Clinical Study Site, Lübeck, Schleswig-Holstein
  - Akero Clinical Study Site, Berlin
- India (17):
  - Akero Clinical Study Site, Hyderabad, Andhra Pradesh
  - Akero Clinical Study Site, Surat, Gujarat
  - Akero Clinical Study Site, Vadodara, Gujarat
  - Akero Clinical Study Site, Mysore, Karnataka
  - Akero Clinical Study Site, Thiruvananthapuram, Kerala
  - Akero Clinical Study Site, Mumbai, Maharashtra
  - Akero Clinical Study Site, Nagpur, Maharashtra
  - Akero Clinical Study Site, Pune, Maharashtra
  - Akero Clinical Study Site, New Delhi, National Capital Territory of Delhi
  - Akero Clinical Study Site, Chandigarh, Punjab
  - Akero Clinical Study Site, Ludhiana, Punjab
  - Akero Clinical Study Site, Jaipur, Rajasthan
  - Akero Clinical Study Site, Coimbatore, Tamil Nadu
  - Akero Clinical Study Site, Hyderabad, Telangana
  - Akero Clinical Study Site, Varanasi, Uttar Pradesh
  - Akero Clinical Study Site, Rishikesh, Uttarakhand
  - Akero Clinical Study Site, Kolkata, West Bengal
- Israel (8):
  - Akero Clinical Study Site, Petah Tikva, Central District
  - Akero Clinical Study Site, Ramat Gan, Central District
  - Akero Clinical Study Site, Haifa, Haifa District
  - Akero Clinical Study Site, Afula, Northern District
  - Akero Clinical Study Site, Nahariya, Northern District
  - Akero Clinical Study Site, Haifa
  - Akero Clinical Study Site, Jerusalem
  - Akero Clinical Study Site, Tel Aviv
- Italy (9):
  - Akero Clinical Study Site, Foggia, Apulia
  - Akero Clinical Study Site, San Giovanni Rotondo, Foggia
  - Akero Clinical Study Site, Rozzano, Milan
  - Akero Clinical Study Site, Torino, Turin
  - Akero Clinical Study Site, Bologna
  - Akero Clinical Study Site, Messina
  - Akero Clinical Study Site, Milan
  - Akero Clinical Study Site, Modena
  - Akero Clinical Study Site, Novara
- Mexico (5):
  - Akero Clinical Study Site, Guadalajara, Jalisco
  - Akero Clinical Study Site, Cuauhtémoc, Mexico City
  - Akero Clinical Study Site, Mexico City, Mexico City
  - Akero Clinical Study Site, Mérida, Yucatán
  - Akero Clinical Study Site, Benito Juárez
- Poland (7):
  - Akero Clinical Study Site, Poznan, Greater Poland Voivodeship
  - Akero Clinical Study Site, Krakow, Lesser Poland Voivodeship
  - Akero Clinical Study Site, Wroclaw, Lower Silesian Voivodeship
  - Akero Clinical Study Site, Lodz, Lódzkie
  - Akero Clinical Study Site, Warsaw, Masovian Voivodeship
  - Akero Clinical Study Site, Częstochowa, Silesian Voivodeship
  - Akero Clinical Study Site, Katowice, Silesian Voivodeship
- Puerto Rico (3):
  - Akero Clinical Study Site, Manatí
  - Akero Clinical Study Site, Mayagüez
  - Akero Clinical Study Site, San Juan
- South Korea (6):
  - Akero Clinical Study Site, Daegu, Daegu Gwang'yeogsi [Taegu-Kwangyokshi]
  - Akero Clinical Study Site, Incheon, Gyeonggi-do
  - Akero Clinical Study Site, Goyang-si, Gyeonggido
  - Akero Clinical Study Site, Daegu, Gyeongsangbugdo [Kyongsangbuk-do]
  - Akero Clinical Study Site, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Akero Clinical Study Site, Seoul, Seoul Teugbyeolsi
- Spain (7):
  - Akero Clinical Study Site, Sabadell, Barcelona
  - Akero Clinical Study Site, Santander, Cantabria
  - Akero Clinical Study Site, Majadahonda, Madrid
  - Akero Clinical Study Site, Barcelona
  - Akero Clinical Study Site, Madrid
  - Akero Clinical Study Site, Seville
  - Akero Clinical Study Site, Valencia
- Switzerland (4):
  - Akero Clinical Study Site, Lugano, Canton Ticino
  - Akero Clinical Study Site, Bern
  - Akero Clinical Study Site, Sankt Gallen
  - Akero Clinical Study Site, Zurich
- Turkey (Türkiye) (3):
  - Akero Clinical Study Site, Ankara
  - Akero Clinical Study Site, Bursa
  - Akero Clinical Study Site, Rize
- United Kingdom (6):
  - Akero Clinical Study Site, London, England
  - Akero Clinical Study Site, Nottingham, England
  - Akero Clinical Study Site, Birmingham
  - Akero Clinical Study Site, London
  - Akero Clinical Study Site, Newcastle upon Tyne
  - Akero Clinical Study Site, Whitechapel